CLINICAL TRIAL: NCT02977871
Title: A Randomized Trial Comparing Bladder Flap Versus Omission of Flap During Cesarean Section of Primiparous Women
Brief Title: Bladder Flap Versus Omission of Flap During Cesarean Section of Primiparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Attending Physician, ObGyn, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1828
Record Dates: First submitted 2016-11-21; First posted 2016-11-30 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Cesarean Section
Keywords: Cesarean section; operating time; bladder; urinary retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Bladder Flap group (No Intervention): Routine uterine incision performed during cesarean section without incision and dissection of the bladder peritoneum.
- Bladder Flap group (Active Comparator): Routine uterine incision performed during cesarean section with an incision and a dissection of a bladder flap.
  Interventions: Procedure: Bladder flap

INTERVENTIONS:
Procedure: Bladder flap — Performing uterine incision and cesarean section with a bladder flap.
  Arms: Bladder Flap group

SUMMARY:
Cesarean section is the most common surgical procedure performed on women. Over the years minor variations of each surgical step have been introduced, and cesarean sections are not standardized and many different techniques are employed during surgery. Creation of a bladder flap has been an integral surgical step of the cesarean section for many years. The role of the bladder flap and its usefulness in cesarean section is not known well. Further, in some cases the bladder flap is omitted during cesarean section. The aim of the current study is to compare operating time and postoperative urinary symptoms in cesarean sections using either bladder flap or omission of flap.

DETAILED DESCRIPTION:
Cesarean section is the most common surgical procedure performed on women. The main aspects of the surgical approach to low-transverse cesarean delivery have not changed much since1926. Over the years minor variations of each surgical step have been introduced, and cesarean sections are not standardized and many different techniques are employed during surgery. Creation of a bladder flap has been an integral surgical step of the cesarean section for many years. The evidence on the role of the bladder flap and its usefulness in cesarean section is very limited. In emergent cesarean sections where rapid delivery is the main goal, the bladder flap is usually omitted. Literature about the usefulness of a bladder flap is limited and more randomized studies are needed. Most of the study outcomes were focusing operating time however, the investigator in the current study additional focused on postoperative urinary symptoms and dynamics. The aim of the current study is to compare operating time and postoperative urinary symptoms in cesarean sections using either bladder flap or omission of flap.

ELIGIBILITY:
Inclusion Criteria:

* primiparous women >37 weeks without high-risk pregnancy

Exclusion Criteria:

* presence of microbiologically confirmed urinary tract infection before delivery, twin pregnancies, cervical dilatation at admission ≥4 cm, estimated fetal weight>4000 gr, history of previous abdominal surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Total operation time | 1 hour
  Total operation time from skin incision to the end of operation

SECONDARY OUTCOMES:
Estimated blood loss | 1 hour
  Estimated blood loss during surgery will be measured in terms of mL
Bladder injury | up to 48 hour
  Bladder injury during cesarean section will be assessed by the number and percentage of patients who had injury
Urinary retention | up to 48 hour
  Postoperative urinary retention will be measured by number and percentage of patients who develop this complication

CONTACTS AND LOCATIONS:
Overall Officials: Berna Aslan Cetin, MD,ObGyn, Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pelosi MA 2nd, Pelosi MA 3rd. Risk factors for bladder injury during cesarean delivery. Obstet Gynecol. 2005 Apr;105(4):900; author reply 901. doi: 10.1097/01.AOG.0000158756.29999.0a. No abstract available. PMID 15802429
- [Result] Wood RM, Simon H, Oz AU. Pelosi-type vs. traditional cesarean delivery. A prospective comparison. J Reprod Med. 1999 Sep;44(9):788-95. PMID 10509303
- [Result] Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery. Am J Obstet Gynecol. 2005 Nov;193(5):1607-17. doi: 10.1016/j.ajog.2005.03.063. PMID 16260200
- [Result] Mahajan NN. Justifying formation of bladder flap at cesarean section? Arch Gynecol Obstet. 2009 Jun;279(6):853-5. doi: 10.1007/s00404-008-0838-6. Epub 2008 Nov 19. PMID 19018545
- [Result] O'Neill HA, Egan G, Walsh CA, Cotter AM, Walsh SR. Omission of the bladder flap at caesarean section reduces delivery time without increased morbidity: a meta-analysis of randomised controlled trials. Eur J Obstet Gynecol Reprod Biol. 2014 Mar;174:20-6. doi: 10.1016/j.ejogrb.2013.12.020. Epub 2013 Dec 22. PMID 24411951
- [Result] Tuuli MG, Odibo AO, Fogertey P, Roehl K, Stamilio D, Macones GA. Utility of the bladder flap at cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2012 Apr;119(4):815-21. doi: 10.1097/AOG.0b013e31824c0e12. PMID 22395144